CLINICAL TRIAL: NCT03828097
Title: The Effects of a Multi-vitamin Supplement on Mood and Blood Markers in Adult Females Prior to and Following 12 Weeks of Supplementation
Brief Title: The Effects of a Multi-vitamin Supplement in Adult Females
Acronym: MVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Michael Roberts, Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-092 MR 1803
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Health, Subjective

STUDY DESIGN:
Intervention Model Description: Double-blinded, parallel
Who Masked: Participant, Investigator
Masking Description: Pills are in white bottles with unique ID numbers (1-110). Pills are also flavor-matched (mint).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental supplement (Experimental): Participants in this arm will receive two capsules per day containing a total of 1 mg boron, 600 mcg folate, 8 mg iron, 50 mg magnesium, 320 mg omega-3 (DHA+EPA), 8 mcg vitamin B12, 50 mcg vitamin D3, and 7 mg vitamin E
  Interventions: Dietary Supplement: Experimental supplement
- Placebo (Placebo Comparator): Participants in this arm will receive two capsules per day containing safflower oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental supplement — Subjects in both arms will consume two pills daily. Prior to and following 12 weeks of supplementation, participants will arrive to the laboratory following an overnight fast in order to donate blood as well as fill out EuroQoL and POMS questionnaires.
  Arms: Experimental supplement
Dietary Supplement: Placebo — Subjects in both arms will consume two pills daily. Prior to and following 12 weeks of supplementation, participants will arrive to the laboratory following an overnight fast in order to donate blood as well as fill out EuroQoL and POMS questionnaires.
  Arms: Placebo

SUMMARY:
The investigators are examining how the daily consumption of a multi-vitamin/mineral supplement affects the following variables in 21-40 year old women:

1. blood levels of various micronutrients (assessed from blood draws using mass spectrometry-based assays)
2. blood cell gene expression patterns (assessed from blood draws and real-time PCR assays)
3. mood (assessed via questionnaires) Blood and questionnaires will be collected prior to supplementation, and 12 weeks into supplementation.

DETAILED DESCRIPTION:
The investigators are testing the efficacy of a multi-vitamin/mineral/omega-3 complex on psychological and physiological measures in pre-menopausal women (21-40 years old) over a 12-week period.

This study will be a double-blinded, placebo-controlled intervention. Briefly, subjects will be screened for inclusion criteria. Eligible subjects will then undergo a pre-testing battery (i.e., T1) and will then be randomly assigned to one of two groups including:

1. Experimental group (anticipated n=50)
2. Control group (anticipated n=50) Subjects will then consume 2 capsules per day for 12 weeks and perform a post-testing battery (i.e., T2) that includes tests performed during the pre-testing battery.

Main outcome (dependent) variables between treatments will include:

1. blood levels of various micronutrients (assessed from blood draws using mass spectrometry-based assays)
2. blood cell gene expression patterns (assessed from blood draws and real-time PCR assays)
3. mood (assessed via questionnaires) Blood and questionnaires will be collected prior to supplementation, and 12 weeks into supplementation.

Statistics used to assess differences between conditions over time will include two-way repeated measures ANOVAs. When significant group*time interactions are observed, the statistical model will be decomposed using LSD post hoc tests.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be healthy adult women (21-40 years)
2. Subjects must possess a body mass index between 20-30 kg/m2
3. Subjects can be of all demographics, race, and skin types
4. Subjects must have a regular menstrual cycle
5. Subjects must have never have smoked tobacco
6. Subjects must be willing to practice at least one of the following methods of birth control: (1) Total abstinence from sexual intercourse with someone of the opposite sex during the study duration; (2) Sexual intercourse with a vasectomized partner; (3) Contraceptive (oral, parenteral, or transdermal) for at least 3 consecutive months prior to and during the study duration; (4) Use of an intrauterine contraceptive device; (5) Other acceptable forms of birth control (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).
7. Subjects must be able to travel to test site on scheduled dates/times without transportation issues.

Exclusion Criteria:

1. Any prescribed medication except for oral contraceptives (not acceptable if oral contraceptives are used to disrupt normal/monthly menstrual cycle) - includes recent antibiotic and/or oral corticosteroid use
2. Medical history including the following: cardiovascular disease, cancer, coagulopathies, current anemia, epilepsy, thyroid disease, parathyroid diseases, diabetes, hepatitis, brain injuries or other brain-related diseases, depression treated with prescription medications, liver diseases, abnormal lipid metabolism, digestive disorders (Crohn's, pancreatitis, ulcerative colitis), multiple sclerosis, muscular dystrophy, asthma/COPD
3. Anyone incapable of adhering to the study protocol or knowing likelihood of moving away from the study site
4. Known allergies to algal oils, high-oleic sunflower oil, coconuts/coconut oil
5. Pregnant (or become pregnant during the course of the study)
6. Past or active smokers
7. Irregular menstrual cycles or amenorrhea
8. Donated blood within two months prior to study entry, and must not donate blood during the study duration
9. Consumers of alcohol, > 5 drinks of alcohol per week; one drink of alcohol was considered to be 142 mL of standard wine, 340 mL of beer, 35 mL of 80-proof liquor, or 10 mL of pure alcohol
10. Dietary practices: more than one fish meal per week, or daily consumption of more than a Tablespoon of flaxseeds
11. Caffeine-containing beverages are allowable if not excessive (more than the equivalent of 6 cups of coffee daily) and if they do not contain added vitamins; energy drinks or energy capsules containing caffeine are allowable if they have been used routinely
12. Dietary Supplements: those taking multivitamin-mineral (MVM), prenatal vitamins, B vitamins, fish oil, krill oil, flaxseed oil dietary supplements. Meal replacement drinks or powders with 100% or more of the Daily Values for vitamins and minerals are also excluded, but if subjects cease their use they can be admitted into the study.

    *Allowable supplements include calcium with or without Vitamin D (if the Vitamin D does not exceed 400 IU daily), fiber supplements not exceeding recommended doses on product labels, melatonin, niacin, herbal supplements without added vitamins, glucosamine/chondroitin, sports supplements, drinks or powders that do not contain vitamins and minerals (for example: protein powders, creatine, electrolytes, nitric oxide enhancers). Other supplements can be considered on a case-by-case basis.
13. Study subjects must not be in active litigation regarding malpractice, workman's compensation, or disability claims.
14. Study subjects must not be employees (temporary, part-time, full-time, etc.) or a family member of the research staff conducting the study.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals self-identifying as females will be eligible for the study.
Enrollment: 94 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of micronutrients | 12 weeks
  Blood serum will be collected at PRE and POST-intervention and assessed for 25-hydroxycholecalciferol (25OHD), and folate as well as 6 associated metabolites [folic acid, 5-methyltetrahydrofolate (5-MeTHF), 5-formyltetrahydrofolate (5-FoTHF), homocysteine (Hcy), S-adenosylmethionine (SAM) and S-adenosylhomocysteine (SAH)]. Overall changes in these metabolites will be compared to pre-intervention values to determine if the experimental intervention was more effective at increasing one or multiple micronutrient levels in serum.
Red blood cell omega-3 and omega-6 concentrations | 12 weeks
  Red blood cells will be collected at PRE and POST-intervention and assayed for red blood cell omega-3 and omega-6 fatty acid content. Overall changes in these metabolites will be compared to pre-intervention values to determine if the experimental intervention was more effective at altering these fatty acid levels in red blood cells.

SECONDARY OUTCOMES:
Blood red blood cell concentrations | 12 weeks
  Whole blood will be collected at PRE and POST-intervention and assessed using a CBC test. The CBC test provides red concentration. Results from these tests will be compared to reference range values for apparently healthy female individuals.
White blood cell concentrations | 12 weeks
  Whole blood will be collected at PRE and POST-intervention and assessed using a CBC test. The CBC test also provides white blood cell concentration. Results from these tests will be compared to reference range values for apparently healthy female individuals.
Serum cholesterol concentrations | 12 weeks
  Whole blood will be collected at PRE and POST-intervention, and serum will be extracted and assessed using a chem-20 test. The chem-20 test provides serum lipid concentrations (i.e., LDL cholesterol, HDL cholesterol). Results from these tests will be compared to reference range values for apparently healthy female individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Kinesiology, Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osburn SC, Roberson PA, Medler JA, Shake J, Arnold RD, Alamdari N, Bucci LR, Vance A, Sharafi M, Young KC, Roberts MD. Effects of 12-Week Multivitamin and Omega-3 Supplementation on Micronutrient Levels and Red Blood Cell Fatty Acids in Pre-menopausal Women. Front Nutr. 2021 Jul 13;8:610382. doi: 10.3389/fnut.2021.610382. eCollection 2021. PMID 34327207